# **INFORMED CONSENT FORM**

The Effect of Guided İmagery Applied Before and After Surgery on Surgical Anxiety, Pain and Analgesic Consumption in Patients Undergoing Total Joint Arthroplasty: A Randomized Controlled Trial

#### INFORMED CONSENT FORM

#### PLEASE TAKE THE TIME TO READ THIS DOCUMENT CAREFULLY

We invite you to participate in the research titled **"The Effect of Guided İmagery Applied Before and After Surgery on Surgical Anxiety, Pain and Analgesic Consumption in Patients Undergoing Total Joint Arthroplasty: A Randomized Controlled Trial,"** conducted by Büşra ERGEN TURAN under the supervision of Assoc. Prof. Dr. Gülay YAZICI. Before deciding or not to participate in this study, you need to know why and how the study will be conducted. Therefore, it is very important that you read and understand this form. If there is anything you do understand or that is unclear to you, or if you would like more information, please ask us.

Participationin this study is entirely <u>voluntary</u>. You have the right to <u>decline</u> to participate in the study or to withdraw from it at any time after joining. <u>Your response to the study will be interpreted as your consent to participate in the research.</u> When answering the questions <u>on the forms</u> provided to you, do not be under any pressure or persuasion from anyone. The information obtained from these forms will be used solely for research purposes.

### 1. Information Regarding the Research:

Research Objective: To examine the effect of guided imagery applied before surgery on anxiety in patients undergoing total joint arthroplasty, and the effect of guided imagery applied after surgery on pain intensity and analgesic consumption.

Research Content: Participants will be asked to complete an Informed Patient Consent Form, a Surgery-Specific Anxiety Scale, a Numerical Rating Scale, and an Analgesic Consumption Tracking Form created for the purposes of the study.

Reason for the Research: [] Scientific research [x] Thesis study

Expected Duration of Research Application (approximately in minutes and/or hours): 60-70 minutes

Expected Number of Participants/Volunteers to Participate in the Research: 128

Location(s) where the Research will be Conducted: Zonguldak Atatürk State Hospital

## 2. Study Participation Consent:

I have read the information above, which must be provided to the participant/volunteer prior to the study, and I fully understand the scope and purpose of the study I am being asked to participate in, as well as the responsibilities that fall upon me as a volunteer. Written and verbal explanations about the study were provided by the researcher named below, I had the opportunity to ask questions and discuss, and I received satisfactory answers. The potential risks and benefits of the study were also explained to me verbally. I understand that I can withdraw from this study at any time and for any reason without having to give a reason, and that I will not face any negative consequences if I do so.

Under these conditions, I voluntarily agree to participate in the study without any pressure or coercion.

| Participant (in their own handwriting) |
|----------------------------------------------------------|
| Name-Surname: |
| Signature: |
| (If applicable) For those under guardianship or custody: |
| Parent or Guardian's (in their own handwriting) |
| Name- |
| Surname: |
| Signature: |

Researcher's Name and Surname: Büşra ERGEN TURAN Signature: